CLINICAL TRIAL: NCT07108426
Title: Evaluation of the Impact of In-Person and Telemedicine-Based Medical Education on Diabetes Care and Outcomes in Hospitalized Patients
Brief Title: Medical Education to Improve Diabetes Care and Outcomes in Hospitalized Patients
Acronym: LELOHG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of Pelotas (Other)
Collaborators: Federal University of Health Science of Porto Alegre (Other); Universidade Federal do Rio Grande (FURG) (Other); Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Jivago da Fonseca Lopes, Principal Investigator, Endocrinologist, Catholic University of Pelotas, Catholic University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 84125324.4.1001.5335
Record Dates: First submitted 2025-07-19; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Diabete Type 2; Hyperglycemic Therapy; Medical Education; Telemedecine
Keywords: diabetes mellitus; telemedicine; medical education; hospital hyperglycemia; insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This is a multicenter, open-label, parallel-group randomized clinical trial designed to assess the impact of a structured medical education program on physicians' knowledge and hospital outcomes in patients with diabetes. Internal medicine resident teams from four Brazilian university hospitals were randomized to either an intervention group, which received a virtual class and 30-day follow-up via WhatsApp®, or a control group with usual practice. Outcomes include improvement in medical knowledge, quality of diabetes-related prescriptions, glycemic control, hospital length of stay, and readmission rates.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine Education Group (Experimental): Internal medicine residents in this group will receive a 30-minute online theoretical class on hospital hyperglycemia, taught by hospital-based endocrinologists. After the class, for 30 days, participants will be included in a continuing medical education group via the WhatsApp® application, where they will receive short educational videos and supporting materials related to diabetes and inpatient glycemic control.
  Interventions: Behavioral: Educational Intervention via Telemedicine
- Routine Clinical Practice Group (No Intervention): Internal medicine residents in this group will not receive any theoretical class or continuing education intervention. They will continue their standard clinical duties and usual care practices during the study period, without additional materials or support related to inpatient diabetes management.

INTERVENTIONS:
Behavioral: Educational Intervention via Telemedicine — A structured educational program delivered remotely through WhatsApp®, including a 30-minute online lecture and daily dissemination of educational content (videos, texts, and practical guidance) on hospital hyperglycemia and glycemic management strategies.
  Arms: Telemedicine Education Group

SUMMARY:
This clinical trial aims to evaluate whether a structured medical education strategy can improve the quality of care provided to hospitalized patients with diabetes or hyperglycemia. Internal medicine residents from four university hospitals in southern Brazil are assigned to two groups: an intervention group receiving a 30-minute online lecture and 30 days of educational follow-up via WhatsApp®, and a control group receiving no additional training.

The primary goal is to assess changes in physicians' knowledge about inpatient glycemic control. Secondary goals include evaluating the quality of insulin prescriptions, rates of hyperglycemia and hypoglycemia, and hospital length of stay.

DETAILED DESCRIPTION:
Hospital hyperglycemia is associated with increased morbidity, length of stay, and hospital costs, especially when not properly managed. Many internal medicine teams lack adequate training on glycemic control in hospitalized patients, and guidelines are not consistently followed in clinical practice.

This multicenter, randomized, open-label trial is designed to evaluate whether a telemedicine-based educational intervention can improve medical knowledge and clinical management of inpatient hyperglycemia. Internal medicine residents from four university hospitals in southern Brazil are randomized by clinical team into two groups: one receives a 30-minute online class and continued support via WhatsApp® for 30 days; the control group receives no intervention.

Medical knowledge is assessed using a validated questionnaire before and after the intervention. Secondary outcomes include the appropriateness of glycemic monitoring and insulin prescriptions, frequency of hyper- and hypoglycemia and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Internal medicine residents from clinical teams at the participating university hospitals in southern Brazil.
* Residents assigned to clinical teams during the intervention month.
* Provided informed consent to participate in the study.

Exclusion Criteria:

* Residents on vacation during the intervention month.
* Residents from teams supervised by endocrinologists.
* Refusal to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Improvement in medical knowledge regarding inpatient hyperglycemia | Baseline and 30 days post-intervention
  Medical knowledge will be assessed using a structured and validated questionnaire on hospital hyperglycemia and diabetes, administered before and 30 days after the intervention. The questionnaire includes multiple-choice clinical case scenarios related to glycemic monitoring, insulin use, treatment errors, and glycemic targets.

SECONDARY OUTCOMES:
Occurrence of hyperglycemia | Last 5 days of hospitalization during the 30-day intervention period
  Percentage of capillary glucose (CG) readings >180 mg/dL during the last 5 days of hospitalization.
Quality of insulin prescription | Last 5 days of hospitalization during the 30-day intervention period
  Proportion of prescriptions that include appropriate insulin regimens (e.g., basal or basal-bolus) versus sliding-scale insulin alone.
Occurrence of hypoglycemia | Last 5 days of hospitalization during the 30-day intervention period
  Percentage of CG readings <70 mg/dL during the last 5 days of hospitalization.
Time in glycemic target range | Last 5 days of hospitalization during the 30-day intervention period
  Percentage of CG readings within the 70-180 mg/dL range during the last 5 days of hospitalization.
Glycated hemoglobin ordered at hospital admission | During the 30-day intervention period
  Proportion of patients for whom glycated hemoglobin (HbA1c) was ordered at admission.
Length of hospital stay | During the 30-day intervention period
  Duration in days from hospital admission to discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Pelotas, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy concerns and lack of participant consent for external data sharing.

REFERENCES:
- [Background] Lopes JDF, Andrade PDR, Borges MT, Krause MC, Simi MOS, Bohlke M, Weinert LS. Medical education on hospital hyperglycemia improving knowledge and outcomes. Arch Endocrinol Metab. 2024 Feb 19;68:e230003. doi: 10.20945/2359-4292-2023-0003. eCollection 2024. PMID 39420910
- [Background] Faruque LI, Wiebe N, Ehteshami-Afshar A, Liu Y, Dianati-Maleki N, Hemmelgarn BR, Manns BJ, Tonelli M; Alberta Kidney Disease Network. Effect of telemedicine on glycated hemoglobin in diabetes: a systematic review and meta-analysis of randomized trials. CMAJ. 2017 Mar 6;189(9):E341-E364. doi: 10.1503/cmaj.150885. Epub 2016 Oct 31. PMID 27799615
- [Background] Mendez CE, Umpierrez GE. Pharmacotherapy for Hyperglycemia in Noncritically Ill Hospitalized Patients. Diabetes Spectr. 2014 Aug;27(3):180-8. doi: 10.2337/diaspect.27.3.180. PMID 26246777
- [Background] Umpierrez GE, Reyes D, Smiley D, Hermayer K, Khan A, Olson DE, Pasquel F, Jacobs S, Newton C, Peng L, Fonseca V. Hospital discharge algorithm based on admission HbA1c for the management of patients with type 2 diabetes. Diabetes Care. 2014 Nov;37(11):2934-9. doi: 10.2337/dc14-0479. Epub 2014 Aug 28. PMID 25168125
- [Background] Horton WB, Law S, Darji M, Conaway MR, Akbashev MY, Kubiak NT, Kirby JL, Thigpen SC. A MULTICENTER STUDY EVALUATING PERCEPTIONS AND KNOWLEDGE OF INPATIENT GLYCEMIC CONTROL AMONG RESIDENT PHYSICIANS: ANALYZING THEMES TO INFORM AND IMPROVE CARE. Endocr Pract. 2019 Dec;25(12):1295-1303. doi: 10.4158/EP-2019-0299. Epub 2019 Aug 14. PMID 31412227
- [Background] Wu EQ, Zhou S, Yu A, Lu M, Sharma H, Gill J, Graf T. Outcomes associated with insulin therapy disruption after hospital discharge among patients with type 2 diabetes mellitus who had used insulin before and during hospitalization. Endocr Pract. 2012 Sep-Oct;18(5):651-9. doi: 10.4158/EP11314.OR. PMID 22440990
- [Background] Bansal V, Mottalib A, Pawar TK, Abbasakoor N, Chuang E, Chaudhry A, Sakr M, Gabbay RA, Hamdy O. Inpatient diabetes management by specialized diabetes team versus primary service team in non-critical care units: impact on 30-day readmission rate and hospital cost. BMJ Open Diabetes Res Care. 2018 Apr 5;6(1):e000460. doi: 10.1136/bmjdrc-2017-000460. eCollection 2018. PMID 29657719
- [Background] Rubin DJ. Hospital readmission of patients with diabetes. Curr Diab Rep. 2015 Apr;15(4):17. doi: 10.1007/s11892-015-0584-7. PMID 25712258
- [Background] Moghissi ES, Korytkowski MT, DiNardo M, Einhorn D, Hellman R, Hirsch IB, Inzucchi SE, Ismail-Beigi F, Kirkman MS, Umpierrez GE; American Association of Clinical Endocrinologists; American Diabetes Association. American Association of Clinical Endocrinologists and American Diabetes Association consensus statement on inpatient glycemic control. Diabetes Care. 2009 Jun;32(6):1119-31. doi: 10.2337/dc09-9029. Epub 2009 May 8. No abstract available. PMID 19429873

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-31): https://cdn.clinicaltrials.gov/large-docs/26/NCT07108426/Prot_SAP_000.pdf